CLINICAL TRIAL: NCT03658031
Title: Effect of Dapagliflozin on the Progression From Prediabetes to T2DM in Subjects With Myocardial Infarction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRGC-04-SI-17-117
Record Dates: First submitted 2018-07-22; First posted 2018-09-05 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-07

CONDITIONS: PreDiabetes; Myocardial Infarction; T2DM (Type 2 Diabetes Mellitus); CVD
MeSH Terms: conditions — Prediabetic State; Myocardial Infarction; Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: After completing baseline measurements, subjects will be randomized to receive in a double blind fashion dapaglfilozin (10 mg/day) or placebo. The drug will be administered each morning before breakfast.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10mg per/day in prediabetes cases with MI before breakfast
  Interventions: Drug: Dapagliflozin 10mg
- Placebo (No Intervention): Antiplatelet, ACEI and Betablockers

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10 mg administered each morning before breakfast
  Arms: Dapagliflozin

SUMMARY:
It is hypothesize that, because dapagliflozin will reverse the metabolic defects responsible for the development of prediabetes (i.e. insulin resistance and beta cell dysfunction) and progression from prediabetes to T2DM (beta cell dysfunction) and will cause weight loss, it will markedly reduce the progression from prediabetes to T2DM and reverse glucose tolerance to NGT in patients with prediabetes experiencing acute myocardial infarction. Further, it is hypothesized that the hemodynamic actions of dapagliflzoin will exert cardiovascular benefit in subjects with prediabetes and acute MI by reducing cardiac remodeling, preserve LV function and decrease the risk of development of heart failure and hospitalization for heart failure.

Hence, aim to examine the impact of SGLT2 inhibitor on T2DM and cardiovascular risk in patients with prediabetes and cardiovascular disease.

The primary objective of the study is to examine the effect of dapagliflozin (10 mg) on the progression from prediabetes to T2DM in patients with prediabetes who experience acute myocardial infarction (MI). A secondary objective is to examine the effect of dapagliflozin on a composite of CV outcome including incidence and hospitalization for heart failure in patients with prediabetes with acute MI. Other secondary outcome is the change from baseline to end of study in LD systolic and diastolic function.

DETAILED DESCRIPTION:
The term prediabetes has been coined to describe an intermediate stage in the transition in glucose tolerance from normal glucose tolerance to overt diabetes. According to the ADA criteria, prediabetes include subjects with impaired fasting glucose (FPG=100-125 mg/dl) and/or impaired glucose tolerance (IGT, 2h-hour plasma glucose after 75 glucose load=140-199 mg/dl). Subjects with prediabetes manifest greater risk of progression to T2DM. The annual conversion rate from prediabetes (IFG/IGT) to T2DM varies among various ethnic groups and ranges between 7-15% . The worldwide estimated prevalence of prediabetes is 25-30% of adult population. The high prevalence of prediabetes and the high rate of progression from prediabetes to T2DM is the principal factor which fuels the worldwide diabetes epidemic.

The strong association between T2DM and risk of cardiovascular disease (CVD) is very well established. T2DM patients without established CVD manifest similar risk of acute myocardial infarction (MI) and death to non-diabetic patients with established CVD . Many epidemiologic studies have demonstrated that the close association between CVD risk and glucose intolerance extends to the prediabetic range. Thus, subjects with prediabetes manifest greater CVD risk than NGT. Since the deterioration in glucose tolerance from NGT, to prediabetes and T2DM is a continuum, the greater risk of CVD in subjects with prediabetes is no surprise. Indeed, numerous studies have documented progressive increase in CVD risk with the increase in the 2-hour plasma glucose concentration. In a meta analysis of 20 studies which included 95,783 patients followed for a mean of 12.4 years, an exponential correlation between CV risk and 2-hour plasma glucose concentration existed, and this relationship extended to the NGT range of 2-hour plasma glucose concentration. When patients were dichotomized based upon the 2h plasma glucose concentration to NGT (2h PG<140 mg/dl) and IGT (2h PG=140-199 mg/dl), IGT subjects consistently manifested greater risk of CVD. The increase in CVD risk in IGT subjects varied in different ethnic groups and ranged from 25-122%. These results collectively suggest a strong relationship between T2DM, prediabetes and CVD risk.

Study Aims and Goals:

The primary aim of the study is to examine the impact of SGLT2 inhibitor on T2DM and cardiovascular risk in patients with prediabetes and cardiovascular disease.

Objectives of this study:

The primary objective of the study is to examine the effect of dapagliflozin (10 mg) on the progression from prediabetes to T2DM in patients with prediabetes who experience acute myocardial infarction (MI). A secondary objective is to examine the effect of dapagliflozin on a composite of CV outcome including incidence and hospitalization for heart failure in patients with prediabetes with acute MI. Other secondary outcome is the change from baseline to end of study in LD systolic and diastolic function.

Study design and methodology:

Patient screening: Subjects admitted to the Heart Hospital with the diagnosis of acute myocardial infarction (Acute MI) will be screened with HbA1c and 75-grams OGTT on the day of discharge. Subjects who will fulfill the following criteria: (1) HbA1c=5.7-6.4%; (2) FPG=100-125 mg/dl or; (3) 2-hour plasma glucose concentration =140-199 mg/dl, will be invited for a repeat OGTT at 4 weeks after MI. Subjects who experienced myocardial infarction in the preceding 4 week but were not screened on discharge also will be allowed to receive an OGTT at 4 weeks after MI. Subjects who fulfilled the criteria of prediabetes on screening but their coronary disease requires surgical revascularization will receive a repeat OGTT at 4 weeks after completing the surgical procedure.

Only subjects who have prediabetes (IFG and/or IGT) according to ADA criteria on the repeat OGTT (at 4 weeks) will be invited to participate in the study.

This study design ensures that elevated FPG and/or 2-hour plasma glucose concentration during the OGTT reflects a genuine prediabetic state, not stress induced hyperglycemia following the acute MI.

576 screen-positive patients (with prediabetes plus acute MI) will comprise the study population. Other than prediabetes and coronary artery disease, subjects must be in good general health as determined by medical history, physical examination, blood chemistries, CBC, TSH, T4, lipid profile, HbA1c, urinanalysis, and EKG. Only subjects whose body weight has been stable (± 4 lbs) over the preceding three months and who do not participate in an excessively heavy exercise program will be included in the study. There will no limitation of LVEF for participation in the study.

After completing the repeat OGTT (4 weeks after the coronary event), eligible subjects will receive a measurement of total body fat with bioimpedence and cardiac echocardiography to quantitate systolic and diastolic LV function.

After completing baseline measurements, subjects will be randomized to receive in a double blind fashion dapaglfilozin (10 mg/day) or placebo. The drug will be administered each morning before breakfast.

Subjects will be randomized in a blocks of 4. Subjects in both treatment groups will be matched on mean for age, BMI, LVEF, FPG, and 2-h plasma glucose concentration. They also will be matched for gender and family history of T2DM.

Follow-up visit:

During year 1, subjects will be seen monthly during the first 4 months (4 visits) and every 2 months during the following 8 months (4 visits) by the study nurse coordinator at the CRC in the Heart Hospital. After year 1, subjects will be seen every 3 months. To ensure compliance and perform a brief interim medical history, telephone calls will be made to each participant every 4-6 weeks to reinforce compliance.

During each visit, medical history and physical examination will be performed. Body weight, waist circumference, standing and reclining (after 5 minutes) blood pressure and fasting plasma glucose will be measured. HbA1c will be measured every 3 months. Subjects will be questioned about possible adverse events of study medication, e.g. genital infections, symptoms of hypovolemia, etc. and a pill count will be performed to assess patient's compliance.

The OGTT will be repeated annually. The HbA1c will be measured every 3 months and plasma lipid profile will be measured annually. Plasma LDL cholesterol will be treated with statin to a target <70 mg/dl, and blood pressure will be treated to a target of <130/90 mmHg. All other post MI therapies, e.g. antiplatelet, ACEI, beta blockers etc. will be administered according to guidelines and Heart Hospital policy.

If the FPG (≥ 126 mg/dl during any visit) or 2-h PG (≥ 200 mg/dl during the OGTT) or HbA1c ( 6.5% during any 3 month visit) measured at any follow-up visit indicates the presence of diabetes, the diagnosis will be confirmed with a repeat OGTT (either 2-h PG 200 mg/dl or FPG 126 mg/dl). If diabetes is confirmed in the repeat OGTT, all baseline studies will be repeated and the subject will be referred to the Diabetes Center at Hamad General Hospital for routine care of their diabetes.

In subjects who will not convert to T2DM during the follow-up, all baseline studies will be repeated at month 36, and pharmacotherapy will be discontinued. This will conclude the study and patients will be returned to their Primary Care Physicians for routine patient care.

Subjects will be recruited over 2 years and will be followed for an additional 1 year. Thus, the first subject recruited into the study will be followed for 3 years and the last subject will be followed for 1 year. The mean follow-up will be 2 years. This will allow sufficient time to obtain the required number of events (conversion to T2DM) in the placebo arm (11% per year). Based upon studies with pioglitazone (ACT NOW) and metformin (DPP) and CANOE study, a mean follow-up of ~2 years allows sufficient time to demonstrated a highly significant reduction in IGT conversion to T2DM. This follow-up period also allows sufficient time to detect long term effects of dapagliflozin on LV function. Incidence of T2DM based upon the ADA criteria, Reversion of glucose tolerance on OGTT to NGT, Change from baseline to 3 years in beta cell function and insulin sensitivity measured with OGTT-derived indices, Incidence of a composite CV outcome comprised of: (1) CV death; (2) non-fatal MI; (3) non-fatal stroke; and (4) hospitalization for heart failure (defined as hospitalization >24 hours requiring intravenous diuretic administration) , Change from baseline to 3 year in left ventricular size, systolic and diastolic function will be worked out.

Sample size; data collection methods:

The annual incidence rate of T2DM in IGT subjects receiving placebo in the Diabetes Prevention Program was 11%. Assuming that dapagliflozin will cause 33% reduction in the progression of IGT to T2DM, It is computed that a total of 240 completers in each arm followed for a mean of 2 years provide 90% power to detect 33% reduction in the incidence of T2DM at alpha=0.05. Assuming a total of 20% drop out rate, the sample size is set out 288 subjects in each arm. Thus, a total of 576 subjects will be recruited into the study.

Previous studies from our group have demonstrated that the 1-year rate of hospitalization for heart failure in patients admitted to the Heart Hospital with acute MI is 21% in the first year after MI. Recent clinical trials (EMPA REG (74) and CANVAS (74)) have demonstrated that SGLT2 inhibitors reduce heart failure hospitalization by 38%. Thus, 288 patients with acute MI in each arm provide >90% power to detect 40 reduction in heart failure hospitalization (part of the composite secondary outcome) by dapagliflozin at alpha <0.05.

Echocardiographic diagnosis of Systolic and Diastolic LV function

Echocardiogram will be done prior to enrollment and at the end of follow-up. To assess LV shape and systolic function and determine whether diastolic dysfunction is present, it is adopted the parameters described in the 2016 American Society of Echocardiography and European Association of Cardiovascular Imaging guidelines:

1. E/e>14; the E/e is the ratio of early mitral inflow velocity (E) to mitral annular early diastolic velocity
2. Septale velocity <7 cm/s or laterale velocity <10 cm/s
3. TR velocity >2.8 m/s; this criterion should not be used in patients with significant pulmonary disease.
4. LA maximum volume index >34mL/m2 (should not be applied in athletes, patients with more than mild mitral valve stenosis or regurgitation, or those in atrial fibrillation).

Other measurement will include: left ventricular ejection fraction, left ventricular end-diastolic volume and left ventricular end-systolic volumes, left ventricular mass index and Global longitudinal strain Oral Glucose Tolerance Test (OTT) Patients will report to the CRC in the morning after 10 hours overnight fast. A catheter will be placed in antecubital vein and three baseline blood samples will be drawn. After drawing the baseline samples, subjects will ingest 75 grams glucose in 300 ml solution. Blood samples will be drawn every 15 minutes for the following 2 hours for the measurements of plasma glucose, insulin and C-peptide concentrations.

Data Management and Analysis plan:

The hazard ratio for the primary outcome (conversion from prediabetes to T2DM) will be estimated from the Cox proportional-hazards model and the percent reduction in risk in the intervention group (dapagliflozin versus placebo) will be computed as 100 x (1 - hazard ratio). The cumulative incidence of conversion from prediabetes to T2DM will be estimated with the Kaplan-Meier method. The Hochberg method will be used to determine statistical significance at the p < 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

1. Acute MI according to AHA criteria 4 weeks prior to recruitment
2. eGFR >60 ml/min
3. stable body weight (+2 kg) in the preceding 3 months
4. diagnosis of prediabetes based upon the ADA criteria (FPG=100-125 mg/dl, and/or 2-hour plasma glucose=140-199 mg/dl

Exclusion Criteria:

1. eGFR<60 ml/min
2. T2DM or T1DM according to the ADA criteria
3. Subjects receiving medications known to affect glucose tolerance
4. Pregnancy or lactation
5. Major organ disease like cancer, chronic pulmonary or liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of T2DM | 36 months
  T2DM in Myocardial patients with prediabetes

CONTACTS AND LOCATIONS:
Overall Officials: Jassim Al-Suwaidi, MD, Principal Investigator — Heart Hospital, HMC
Locations (1):
- Heart Hospital, Hamad Medical Coorporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdul-Ghani M, Migahid O, Megahed A, Singh R, Kamal D, DeFronzo RA, Jayyousi A. Insulin secretion predicts the response to therapy with exenatide plus pioglitazone, but not to basal/bolus insulin in poorly controlled T2DM patients: Results from the Qatar study. Diabetes Obes Metab. 2018 Apr;20(4):1075-1079. doi: 10.1111/dom.13189. Epub 2018 Jan 15. PMID 29227578
- [Result] Abdul-Ghani MA, DeFronzo RA. Pathophysiology of prediabetes. Curr Diab Rep. 2009 Jun;9(3):193-9. doi: 10.1007/s11892-009-0032-7. PMID 19490820
- [Result] Genuth S, Alberti KG, Bennett P, Buse J, Defronzo R, Kahn R, Kitzmiller J, Knowler WC, Lebovitz H, Lernmark A, Nathan D, Palmer J, Rizza R, Saudek C, Shaw J, Steffes M, Stern M, Tuomilehto J, Zimmet P; Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Follow-up report on the diagnosis of diabetes mellitus. Diabetes Care. 2003 Nov;26(11):3160-7. doi: 10.2337/diacare.26.11.3160. No abstract available. PMID 14578255
- [Result] Abdul-Ghani MA, Tripathy D, DeFronzo RA. Contributions of beta-cell dysfunction and insulin resistance to the pathogenesis of impaired glucose tolerance and impaired fasting glucose. Diabetes Care. 2006 May;29(5):1130-9. doi: 10.2337/diacare.2951130. PMID 16644654
- [Result] Dankner R, Abdul-Ghani MA, Gerber Y, Chetrit A, Wainstein J, Raz I. Predicting the 20-year diabetes incidence rate. Diabetes Metab Res Rev. 2007 Oct;23(7):551-8. doi: 10.1002/dmrr.728. PMID 17315136
- [Result] Lambers Heerspink HJ, de Zeeuw D, Wie L, Leslie B, List J. Dapagliflozin a glucose-regulating drug with diuretic properties in subjects with type 2 diabetes. Diabetes Obes Metab. 2013 Sep;15(9):853-62. doi: 10.1111/dom.12127. Epub 2013 Jun 5. PMID 23668478
- [Result] Al-Lawati JA, Sulaiman KJ, Al-Zakwani I, Alsheikh-Ali AA, Panduranga P, Al-Habib KF, Al-Suwaidi J, Al-Mahmeed W, Al-Faleh H, El-Asfar A, Al-Motarreb A, Ridha M, Bulbanat B, Al-Jarallah M, Bazargani N, Asaad N, Amin H. Systolic Blood Pressure on Admission and Mortality in Patients Hospitalized With Acute Heart Failure: Observations From the Gulf Acute Heart Failure Registry. Angiology. 2017 Aug;68(7):584-591. doi: 10.1177/0003319716672525. Epub 2016 Oct 7. PMID 27814267
- [Result] Sulaiman K, Panduranga P, Al-Zakwani I, Alsheikh-Ali AA, AlHabib KF, Al-Suwaidi J, Al-Mahmeed W, AlFaleh H, Elasfar A, Al-Motarreb A, Ridha M, Bulbanat B, Al-Jarallah M, Bazargani N, Asaad N, Amin H. Clinical characteristics, management, and outcomes of acute heart failure patients: observations from the Gulf acute heart failure registry (Gulf CARE). Eur J Heart Fail. 2015 Apr;17(4):374-84. doi: 10.1002/ejhf.245. Epub 2015 Mar 4. PMID 25739882
- [Result] Abdul-Ghani M, Migahid O, Megahed A, Adams J, Triplitt C, DeFronzo RA, Zirie M, Jayyousi A. Erratum. Combination Therapy With Exenatide Plus Pioglitazone Versus Basal/Bolus Insulin in Patients With Poorly Controlled Type 2 Diabetes on Sulfonylurea Plus Metformin: The Qatar Study. Diabetes Care 2017;40:325-331. Diabetes Care. 2017 Aug;40(8):1134. doi: 10.2337/dc17-er08d. Epub 2017 Jun 14. No abstract available. PMID 28615237
- [Result] Abdul-Ghani M, Migahid O, Megahed A, Adams J, Triplitt C, DeFronzo RA, Zirie M, Jayyousi A. Combination Therapy With Exenatide Plus Pioglitazone Versus Basal/Bolus Insulin in Patients With Poorly Controlled Type 2 Diabetes on Sulfonylurea Plus Metformin: The Qatar Study. Diabetes Care. 2017 Mar;40(3):325-331. doi: 10.2337/dc16-1738. Epub 2017 Jan 17. PMID 28096223
- [Result] Abdul-Ghani MA, Puckett C, Triplitt C, Maggs D, Adams J, Cersosimo E, DeFronzo RA. Initial combination therapy with metformin, pioglitazone and exenatide is more effective than sequential add-on therapy in subjects with new-onset diabetes. Results from the Efficacy and Durability of Initial Combination Therapy for Type 2 Diabetes (EDICT): a randomized trial. Diabetes Obes Metab. 2015 Mar;17(3):268-75. doi: 10.1111/dom.12417. Epub 2015 Jan 7. PMID 25425451
- [Result] Verma S, Garg A, Yan AT, Gupta AK, Al-Omran M, Sabongui A, Teoh H, Mazer CD, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass and Diastolic Function in Individuals With Diabetes: An Important Clue to the EMPA-REG OUTCOME Trial? Diabetes Care. 2016 Dec;39(12):e212-e213. doi: 10.2337/dc16-1312. Epub 2016 Sep 27. No abstract available. PMID 27679584
- [Result] Oliva RV, Bakris GL. Blood pressure effects of sodium-glucose co-transport 2 (SGLT2) inhibitors. J Am Soc Hypertens. 2014 May;8(5):330-9. doi: 10.1016/j.jash.2014.02.003. Epub 2014 Feb 12. PMID 24631482
- [Result] Al-Jobori H, Daniele G, Cersosimo E, Triplitt C, Mehta R, Norton L, DeFronzo RA, Abdul-Ghani M. Empagliflozin and Kinetics of Renal Glucose Transport in Healthy Individuals and Individuals With Type 2 Diabetes. Diabetes. 2017 Jul;66(7):1999-2006. doi: 10.2337/db17-0100. Epub 2017 Apr 20. PMID 28428225